CLINICAL TRIAL: NCT03693495
Title: A Prospective Multi-Centre Study of the Performance of Ellume·Lab Group A Strep Test Versus Culture for the Rapid Detection of Group A Streptococcus in Participants With Acute Pharyngitis
Brief Title: Performance of Ellume·Lab Group A Strep Test Versus Culture for the Rapid Detection of Group A Streptococcus in Participants With Acute Pharyngitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was cancelled before enrollment for reasons not related to safety and performance.
Sponsor: Ellume Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E-GAS-NZ-1807
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Group A Streptococcal Infection
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ellume·lab Group A Streptococcus Test (Experimental): ellume·lab Group A Streptococcus Test
  Pharyngeal samples from participants will be tested with:
  ellume.lab Group A Streptococcus Test; Polymerase Chain Reaction (PCR) and bacterial culture.
  Interventions: Diagnostic Test: ellume·lab Group A Streptococcus Test; Diagnostic Test: Bacterial Culture; Diagnostic Test: Polymerase Chain Reaction (PCR)

INTERVENTIONS:
Diagnostic Test: ellume·lab Group A Streptococcus Test — ellume.lab Group A Streptococcus Test is a rapid diagnostic test intended to be used as an aid in the diagnosis of Group A Streptococcus in symptomatic participants. The sample type used is a throat swab.
Diagnostic Test: Bacterial Culture — Pharyngeal swab is collected from participant and this specimen is inoculated into 5% sheep blood agar plates. Beta-haemolytic colonies are isolated, followed by latex agglutination test.
Diagnostic Test: Polymerase Chain Reaction (PCR) — Polymerase Chain Reaction (PCR) is a molecular diagnostic technique for the detection and identification of Group A Streptococcus, both for clinical samples and isolates. Polymerase Chain Reaction (PCR) allows template bacterial RNA to be reverse transcribed producing complementary DNA (cDNA) which can then be amplified and detected.

SUMMARY:
Participants who meet the eligibility criteria and who consent to participation or whose parents/legal guardian consent to their participation, will be enrolled in the study for a period of up to 14 days. Enrolment visit (Day 1) assessments for all participants will include the collection of throat swabs, testing by staff at the site using the ellume·lab Group A Strep Test and testing for Group A Streptococcus by a central laboratory using bacterial culture and polymerase chain reaction (PCR). All participants will be followed up with a phone assessment of adverse events between Days 2-14.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants aged 3 years of age or older
* Must currently be presenting with symptoms characteristic of pharyngitis, possibly Group A Strep, including:

  * Acute onset of sore throat;
  * Fever ≥ 37.8° C (100° F) at presentation or history or parent/guardian-reported history of fever ≥ 37.8° C or feeling feverish within 24 hours of presentation and;
  * At least one of the following:

    * Red and swollen/inflamed tonsils (or fossae);
    * Pharyngeal or tonsillar exudate; o Cervical lymphadenopathy
* ≤ 14 days from onset of signs and symptoms of pharyngitis
* Parent/legal guardian of Participants < 18 years of age capable and willing to give informed consent
* Participants ≥18 years of age capable and willing to give informed consent

Exclusion Criteria:

* Participants < 3 years of age
* Participants undergoing treatment with antibiotics, or those who have undergone treatment with antibiotics for current episode of pharyngitis
* Currently enrolled in another clinical trial or used any investigational device within 30 days preceding informed consent
* Participants 18 years of age or older unable to understand English and consent to participation
* Parent/legal guardian of Participants < 18 years of age unable to understand English and consent to participation of child
* Prior enrollment in this clinical validation study

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of the ellume·lab Group A Strep Test in detecting Group A Streptococcus in samples collected using a throat swab as compared to bacterial culture | 1 Week
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence intervals
The specificity of the ellume·lab Group A Strep Test in detecting Group A Streptococcus in samples collected using a throat swab as compared to bacterial culture | 1 Week
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence intervals

SECONDARY OUTCOMES:
The sensitivity of the ellume·lab Group A Strep Test in detecting Group A Streptococcus in samples collected using a throat swab as compared to PCR | 1 Week
  Establish sensitivity against a gold standard. Report as a percentage of participants with 96% confidence intervals
The specificity of the ellume·lab Group A Strep Test in detecting Group A Streptococcus in samples collected using a throat swab as compared to PCR | 1 Week
  Establish specificity against a gold standard. Report as a percentage of participants with 96% confidence intervals
Ease of use as assessed by operator questionnaire | 1 Week
  The ease of use questionnaire will provide total number of responses to each question and the percentage of participants selecting each response (on a 5 point Likert scale).

CONTACTS AND LOCATIONS:
Overall Officials: Barnaby H Montgomery, Principal Investigator — Optimal Clinical Trials
Locations (4):
- New Zealand (4):
  - Optimal Clinical Trials, Grafton, Auckland
  - Totara Clinical Research Ltd, New Lynn, Auckland
  - Papamoa Pines Medical Centre, Papamoa, Tauranga
  - Lakeland Clinical Trials, Rotorua

IPD SHARING:
Plan to Share IPD: No